CLINICAL TRIAL: NCT04382443
Title: Oral Colchicine in Argentina (ORCA Trial) for the Prevention of Adverse Events After Percutaneous Coronary Interventions
Brief Title: Oral Colchicine in Argentina to Prevent Restenosis
Acronym: ORCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de estudios en Cardiologia Intervencionista (Other)
Responsible Party: Principal Investigator, Alfredo E Rodriguez, MD, PhD, Centro de estudios en Cardiologia Intervencionista
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CECI-03
Record Dates: First submitted 2020-03-31; First posted 2020-05-11 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Restenosis of Coronary Artery Stent; Atherosclerosis; Acute Coronary Syndrome
Keywords: restenosis; atherosclerosis; acute coronary syndrome; percutaneous coronary intervention; colchicine; inflammation
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Acute Coronary Syndrome; Inflammation | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Colchicine +BMS implantation (Experimental): This group will receive after BMS and Colchicine, at the time of PCI, 0,5 mg twice a day during the first three months after stent implantation
  Interventions: Drug: Colchicine
- Second generation Drug eluting stent (DES) (No Intervention): This group will receive DES at the moment of randomization and will be treated as standard of care.
  All second generation DES should be approved by ANMAT for clinical use.

INTERVENTIONS:
Drug: Colchicine — At the moment of BMS implantation intervention will mean that this group will receive colchicine as described.
  Other Names: BMS+Colchicine
  Arms: Oral Colchicine +BMS implantation

SUMMARY:
The Oral treatment of Colchicine in Argentina (ORCA) trial is a prospective, randomized, multicenter trial to included 450 patients with indication for myocardial revascularization with PCI between a group to be treated with BMS plus oral colchicine (OC) for three months, which should be administered at the time of PCI, these patients they would receive 0.5 mg twice a day per 3 months compared to the other group of patients who will be treated exclusively with last generation of DES.

DETAILED DESCRIPTION:
In a previous randomized comparison oral colchicine plus bare metal stent (BMS) compared to BMS plus placebo in a diabetic High risk for re-stenosis population, OC demonstrate a significant reduction of angiographic and intravascular ultrasound parameters of in-stent restenosis (ISR) after BMS implantation at one year of follow up (Journal of the American College of Cardiology,2013,61,1678-1685), with a clinical indication of target lesion revascularization in 3.6%. In addition previous reported registries from our group with Drug Eluting Stents showed similar amount of reduction in clinical parameters (not angiographic) of restenosis (ERACI III trial, one year TVR in 8.8% with 1st DES design, Rodriguez A et al EuroIntervention 2006,2:53-60 and 4.0% with 2nd generation DES design ERACI IV Cardiac and cardiovascular interventions Journal, 2014 ). Taking in account those numbers the investigators sought to compare differences in overall cost with both revascularization strategies at 1, 2, 3 and 5 years of follow up assuming that safety and efficacy clinical end points would be similar. Cost included in hospital, procedural and resources fees, follow up cost including re-hospitalization driving by target vessel revascularization (TVR) and both spontaneous and TVR myocardial infarction (MI) and medication cost for each revascularization strategies Safety end point will be incidence of major adverse cardiac events (MACE) defined as the composite of death from any cause, MI (peri-procedural and spontaneous at follow up) and ischemic driving TVR.

The study will be considered complete after all subjects have completed the 12-month Primary safety and efficacy endpoint was incidence of target vessel failure (TVF) plus one year overall cost with both strategies.. Additional end points are clinical endpoints measured in-hospital at at follow up period. cardiac death, cardiac death plus MI. spontaneous MI beyond 30 day to 5 years, and stent thrombosis rate (ST) (definite or probable by Academic Research Consortium definitions).

A sub-study of changes in biological markers of inflammation in patients with acute coronary syndrome (ACS) including MI will be analyzed in both groups. For this reason, a measurement of interleukin 6, metalloproteases, adiponectin and Protein C reactive (PCR) will be performed at the time of enrolment and 4 days and a month after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and angiographic

  1. Subject must be at least 18 to 80 years of age.
  2. Subject (or legal guardian) indicates understanding of the trial requirements and the treatment procedures and provides written informed consent before procedures are performed.
  3. Subject is eligible for PCI
  4. Subject has symptomatic coronary artery disease or silent ischemia with objective evidence of ischemia, or acute coronary syndromes, and qualifies for PCI

  6. Subject has a left ventricular ejection fraction (LVEF) > 40 % as measured within 60 days prior to enrollment.

  7. Subject is willing to comply with all protocol-required follow-up evaluations.

  8. Subject has one or more coronary artery stenosis of ≥ 70 % in a coronary artery with visually estimated reference vessel diameter (RVD) ≥2.50 mm.

Exclusion Criteria:

Clinical and angiographic

1. Subject has a known allergy to contrast (that cannot be adequately pre-medicated) and/or the stent system or Colchicine. (e.g., cobalt chromium alloy, stainless steel, all P2Y12 inhibitors, or aspirin)
2. Planned surgery within 30 days after the index procedure
3. Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 36 months.
4. Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.)
5. Planned procedure that may cause non-compliance with the protocol or confound data interpretation.
6. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions

5. Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint, or that, in the opinion of the investigator, may cause non-compliance with the protocol or confound data interpretation.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
MACE | 365 days
  MACE: Was defined as a composite of death, Myocardial infarction (MI) Stroke, stroke and ischemic target vessel revascularization (TVR) Death included cardiac, non- cardiac and non- determined. MI included STEMI with new q waves at the EKG and /or 5 times increase cardiac enzymes elevation for baseline levels. NSTEMI included 5 times enzymes elevation with non- new Q waves.
  TVR included repeat revascularization in the target vessel initially treated driving by new chest pain and / or perfusion ischemic changes at ergometric or perfusion test.

SECONDARY OUTCOMES:
Target lesion failure | 365 days
  Target lesion failure (TLF): TLF was defined as cardiac death, MI and ischemic driving revascularization (TLR) of initially treated lesion.

OTHER OUTCOMES:
Changes C-Reactive Protein (CRP) values | baseline, 4 and 30 days
  Normal values: 0 to 5 mg/L
Changes in Adinopectine values μU/mL | baseline and 30 days
  Normal values in women 4,62±1,57 vs In men 3,93±1,86 μU/mL
Changes in Interleukin 6 values (pg/m) | baseline and 30 days
  Normal values IL-6 (5-15 pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo E Rodriguez, MD, PhD, Study Chair — Centro de estudios en Cardiologia Intervencionista
Locations (2):
- Argentina (2):
  - Sanatorio Otamendi, Ciudad de Buenos Aires, Buenos Aires
  - Sanatorio Las Lomas, San Isidro, Buenos Aires

IPD SHARING:
Plan to Share IPD: Yes
All researchers that want to work with the database must sign a confidentiality form and all legal documents applicable for the time being.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From May 2020 to December 2022
Access Criteria: Researcher with approved HIPPA compliant certificates. Accept to sign confidentiality form. Do not publish content without autorization of the Sponsor or Chair of the trial.

REFERENCES:
- [Background] Correa-Sadouet C, Rodriguez-Granillo AM, Gallardo C, Mieres J, Fontana L, Curotto MV, Wainer P, Allende NG, Fernandez-Pereira C, M Vetulli H, la Hoz RP, Kastrati A, Rodriguez AE; ORCA investigators. Randomized comparison between bare-metal stent plus colchicine versus drug-eluting stent alone in prevention of clinical adverse events after percutaneous coronary intervention. Future Cardiol. 2021 Jul;17(4):539-547. doi: 10.2217/fca-2020-0161. Epub 2020 Nov 11. PMID 33174761
- [Derived] Rodriguez-Granillo AM, Mieres J, Fernandez-Pereira C, Sadouet CC, Milei J, Swieszkowski SP, Stutzbach P, Santaera O, Wainer P, Rokos J, Gallardo C, Cristodulo-Cortez R, Perez de la Hoz R, Kastrati A, Rodriguez AE, On Behalf Of Orca Investigators. Randomized Clinical Trial Comparing Bare-Metal Stents Plus Colchicine Versus Drug-Eluting Stents for Preventing Adverse Cardiac Outcomes: Three-Year Follow-Up Results of the ORal Colchicine in Argentina (ORCA) Trial. J Clin Med. 2025 Apr 22;14(9):2871. doi: 10.3390/jcm14092871. PMID 40363904